CLINICAL TRIAL: NCT01679626
Title: The Effect of Cricoid Pressure and Backward Upward Rightward Pressure on Airway Dimensions - Implications for Airway Management?
Brief Title: Airway Manoeuvers - Implications for Airway Management?
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Ralph Maassen, MD, principal investigator, Catharina Ziekenhuis Eindhoven
Other Study IDs: 2011-06
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Airway Management
Keywords: cricoid pressure (CP); backward upward rightward pressure (BURP); AP-rima distances; Glottic area; Extralaryngeal manoeuvres

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In anesthesia, intubation is a technique used to secure an airway. This technique is not always straightforward. Sometimes it is difficult to place an endotracheal tube. There are two manners of giving pressure to the patients neck, to improve view and facilitate intubation.

The investigators hypothesize that by giving this pressure the effective work area is likely to be smaller. The investigators would like to quantify this effect by measuring the effective work area, using a specially designed computer program.

DETAILED DESCRIPTION:
Cricoid pressure (CP) and the backward-upward-rightward pressure (BURP) manoeuver, are extralaryngeal manoeuvers which are widely applied during endotracheal intubation, respectively offering potential protection against passive gastric regurgitation and improved laryngeal view in emergency airway management.

Their validity in achieving an improvement of the laryngeal view has been questioned.

The objective of this study is to measure the change in mean anterior-posterior rima glottidis (APRIMA) distance and mean area under the vocal cords after backward upward rightward pressure (BURP) and cricoid pressure (CP).

The investigators will measure the APRIMA distances and areas under the vocal cords, using a specially created module in the program DeVIDE. The measurements assessed during BURP and CP will be expressed relative to the measurements when no external pressure is applied.

ELIGIBILITY:
Inclusion Criteria:

- 200 consecutive adult patients scheduled for elective surgery requiring endotracheal intubation

Exclusion Criteria:

* BMI > 35 kg.m-2);
* chronic obstructive pulmonary disease;
* history of difficult intubation;
* mouth opening < 3 cm;
* inadequate neck mobility;
* history of oropharyngeal pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 consecutive adult patients scheduled for elective surgery requiring endotracheal intubation.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, Netherlands